CLINICAL TRIAL: NCT02170571
Title: Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of 150 mg Dabigatran Etexilate p.o. in Patients With Moderate Hepatic Impairment Compared to Subjects With Normal Hepatic Function in a Monocentric, Open, Parallel-group Design
Brief Title: Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of Dabigatran Etexilate in Patients With Moderate Hepatic Impairment Compared to Subjects With Normal Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1160.51
Record Dates: First submitted 2014-06-20; First posted 2014-06-23 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Hepatic Insufficiency
MeSH Terms: conditions — Hepatic Insufficiency | interventions — Dabigatran

ARMS (1):
- Dabigatran etexilate (Experimental)
  Interventions: Drug: Dabigatran etexilate

INTERVENTIONS:
Drug: Dabigatran etexilate

SUMMARY:
Assessment of the effect of moderate liver impairment (Child-Pugh classification B) on the pharmacokinetics and pharmacodynamics of dabigatran after oral administration of dabigatran etexilate. Determination of safety and tolerability of dabigatran upon administration to hepatically impaired patients and healthy subjects (matched pairs)

ELIGIBILITY:
Inclusion Criteria:

* Healthy age-, weight-, and sex-matched subjects determined by results of screening with normal hepatic function (group 1)
* Hepatically impaired subjects determined by results of screening classified as Child-Pugh B (group 2)
* Signed written informed consent in accordance with Good Clinical Practice (GCP) and local legislation
* Age >=18 and <=75 years
* BMI >=18.0 and <=32 kg/m2, at least 45 kg for females
* Creatinine clearance >80 mL/min according to Cockcroft & Gault

Exclusion Criteria:

* Healthy subjects (Group 1) who met any of the following criteria should not be entered into this trial:

  * Any finding of the medical examination (including blood pressure, pulse rate, and electrocardiogram) deviating from normal and of clinical relevance
  * Clinically relevant gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic or hormonal disorders
  * Surgery of gastrointestinal tract (except appendectomy, cholecystectomy, herniotomy)
  * Clinically relevant diseases of the central nervous system
  * Relevant history of orthostatic hypotension, fainting spells or blackouts
  * Evidence of blood dyscrasia, haemorrhagic diathesis, severe thrombocytopenia, cerebrovascular haemorrhage, bleeding tendencies associated with active ulceration or overt bleeding of gastrointestinal, respiratory or genitourinary tract or any disease or condition with haemorrhagic tendencies (e.g. cerebral aneurysm, dissecting aorta, central nervous system (CNS) trauma, retinopathy, nephrolithiasis)
  * Recent or contemplated diagnostic or therapeutic procedures with potential for uncontrollable bleeding (e.g. spinal puncture, lumbar block anaesthesia, surgery of CNS or eye or surgery resulting in large open surfaces) within 14 days before or after drug administration of this clinical trial
  * Chronic or relevant acute infections
  * History of allergy/hypersensitivity (including drug allergy), which is deemed relevant to the trial as judged by the investigator
  * For women with childbearing potential: no reliable contraception (accepted methods are intra-uterine device, hormonal contraceptives, bilateral tubal ligation, hysterectomy, condoms) or pregnancy (known or detected by a positive pregnancy test) or breast feeding period
  * Intake of drugs with a long half-life (> 24 hours) (< 1 month prior to administration or during the trial)
  * Use of any drugs, within 14 days prior to administration or during the trial
  * Participation in another trial with an investigational drug (< 2 months prior to administration or during trial)
  * Drug abuse
  * Blood donation or loss > 400 ml, < 1 month prior to administration or during the trial
  * Excessive physical activities < 5 days prior to administration of study drug or during the trial
  * Clinically relevant laboratory abnormalities
  * Veins unsuited for i.v. puncture and administration of prolonged infusions on either arm (e.g. veins which are difficult to locate, access or puncture, veins with a tendency to rupture during or after puncture, etc.)
* Hepatically impaired subjects (Group 2) who met any of the following criteria should not be entered into this trial:

  * Moderate and severe concurrent renal function impairment (e.g., due to hepato-renal syndrome)
  * Clinically relevant gastrointestinal, respiratory, cardiovascular, metabolic, immunologic or hormonal disorders
  * Surgery of gastrointestinal tract (except appendectomy, cholecystectomy, herniotomy)
  * Clinically relevant diseases of the central nervous system
  * Relevant history of orthostatic hypotension, fainting spells or blackouts
  * Evidence of blood dyscrasia, haemorrhagic diathesis, severe thrombocytopenia, cerebrovascular haemorrhage, bleeding tendencies associated with active ulceration or overt bleeding of gastrointestinal, respiratory or genitourinary tract or any disease or condition with haemorrhagic tendencies (e.g. cerebral aneurysm, dissecting aorta, CNS trauma, retinopathy, nephrolithiasis) considered by the investigator or one of the coinvestigators to be clinically relevant
  * Recent or contemplated diagnostic or therapeutic procedures with potential for uncontrollable bleeding (e.g. spinal puncture, lumbar block anaesthesia, surgery of CNS or eye or surgery resulting in large open surfaces) within 14 days before or after drug administration of this clinical trial
  * History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
  * For women with childbearing potential: no reliable contraception (accepted methods are intra-uterine device, hormonal contraceptives, bilateral tubal ligation, hysterectomy, condoms) or pregnancy (known or detected by a positive pregnancy test) or breast feeding period
  * Use of any drugs which have an influence on the blood clotting within 14 days prior to administration or during the trial
  * Participation in another trial with an investigational drug (< 2 months prior to administration or during trial)
  * Blood donation or loss > 400 ml, < 1 month prior to administration or during the trial
  * Excessive physical activities < 5 days prior to administration of study drug or during the trial
  * Clinically relevant laboratory abnormalities (except for liver function tests according to Child-Pugh classification), constellation of blood clotting parameters according to the judgment of the investigator
  * Veins unsuited for i.v. puncture and administration of prolonged infusions on either arm (e.g. veins which are difficult to locate, access or puncture, veins with a tendency to rupture during or after puncture, etc.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-07; Primary Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
AUC0-infinity (area under the concentration time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 hours
Cmax (maximum concentration of the analyte in plasma) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 hours
CL/F (apparent clearance of the analyte in the plasma after extravascular administration) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 h
concentration-response relationship of dabigatran assessed by analysis of activated partial thromboplastin time (aPTT), ecarin clotting time (ECT) , prothrombin time (PT) expressed as international normalised ratio (INR), and thrombin time (TT) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 h

SECONDARY OUTCOMES:
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 h
AUCt1-t2 (Area under the concentration time curve of the analyte in plasma over the time interval t1 to t2) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 h
tmax (time from dosing to the maximum concentration of the analyte in plasma) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 h
λz ( terminal rate constant in plasma) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 h
t1/2 ( terminal half-life of the analyte in plasma) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 h
MRTpo (mean residence time of the analyte in the body after oral administration) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 h
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 h
Ae0-72 (amount of analyte that is eliminated in urine from the time interval 0 to 72 h) | pre-dose over 12 h from day -1 till day 1 and post-dose from day 1 till day 4 in fractions of 0 - 12, 12 - 24, 24 - 48 and 48 - 72 h
fe0-72 (fraction of administered drug excreted unchanged in urine from time point 0 to 72 h) | pre-dose over 12 h from day -1 till day 1 and post-dose from day 1 till day 4 in fractions of 0 - 12, 12 - 24, 24 - 48 and 48 - 72 h
CLR,0-72 (renal clearance of the analyte in plasma from the time point 0 h until the time point 72 h) | pre-dose over 12 h from day -1 till day 1 and post-dose from day 1 till day 4 in fractions of 0 - 12, 12 - 24, 24 - 48 and 48 - 72 h
Plasma protein binding of dabigatran | before drug administration
Change in pulse rate | up to day 4
Change in systolic and diastolic blood pressure | up to day 4
Change in ECG | up to day 4
Occurrence of adverse events | up to Day 4
Assessment of tolerability by investigator on a four-point scale | up to day 4